CLINICAL TRIAL: NCT04611256
Title: Adjuvant Therapy With Mesenchymal Stem Cells in Patients Diagnosed With COVID-19 in Critical Condition
Brief Title: Mesenchymal Stem Cells in Patients Diagnosed With COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Reg. Lic. Adolfo Lopez Mateos (Other Government)
Collaborators: Instituto de Terapia Celular: ITC (Unknown)
Responsible Party: Principal Investigator, M. Eunice Rodríguez Arellano, MD, Hospital Reg. Lic. Adolfo Lopez Mateos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060I.2020
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: COVID-19; Adjuvant therapy; mesenchymal stem cells; Mexico
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC transfusion (Experimental)
  Interventions: Biological: MSC
- Control (Active Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Biological: MSC — Two intravenous infusion of 1*10E6 adipose tissue derived-MSCs /kg body weight reach
  Arms: MSC transfusion
Drug: Control — Conventional treatment that may include analgesic, anti-inflammatory, antibiotic, steroid, antiplatelet, and anticoagulant.
  Arms: Control

SUMMARY:
The propose of this study is implement adjuvant therapy with adipose tissue derived-mesenchymal stem cells (MSCs) for critical COVID-19 patients admitted to the intensive care unit of the Regional Hospital Lic. Adolfo López Mateos of the Institute for Social Security and Services for State Workers to reduce cytokine storm and contribute to the favorable resolution of respiratory insufficiency and multiple organic failure.

DETAILED DESCRIPTION:
Within the epidemic context of phase 3 that currently exists in Mexico, implementation of new treatments that have shown to be beneficial for patients in a critical state in other countries is an urgent need. Adipose tissue derived-mesenchymal stem cells for could favor the regulation of patient immune system to reduce the proinflammatory state and promoting the regeneration of damaged tissues.

Patients diagnosed COVID-19 and confirmed positive with the virus by PCR, will be treated with two intravenous infusions MSCs on the day 1 (D1) and the day 3 (D3) of the treatment consisting of 1X106/kg each.

We will assess the pulmonary lesion area by chest x-ray or computed axial tomography at baseline and days 2, 3, 5, 10, 15, 20, and 25.

Days to clinical improvement (to be evaluated on days 2, 3, 5, 10, 15, 20, 25), considering temperature and other vital signs measurement, arterial oxygen saturation, blood chemistry (including liver function tests), creatine phosphokinase, C reactive protein, immune cells (CD3+, CD4+, CD8+, CD16+, CD19+, and CD56+ lymphocytes), pro-inflammatory cytokines (IL-1β, IL- 2, TNF-α, ITN-γ, IL-4, IL-6, IL-10), immunoglobulins (IgA, IgG, IgM, and IgE), HLA profile expression, and weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65.
* RT-PCR positive for SARS-CoV-2 (Berlin protocol).
* Moderate to severe acute respiratory insufficiency (100 mmHg <PaO2/FiO2 ≤ 200 mmHg).
* Confirmatory diagnosis of pulmonary injury by chest teleradiography or computed axial t tomography.
* Being under standard therapy for COVID-19.
* Informed consent signed by the patient or a legally acceptable representative (in the case of the legal representative, informed consent could be obtained by a phone call or email with the subsequent written confirmation).

Exclusion Criteria:

* Reserved prognosis (survival expected by the physician of fewer than three days).
* Being under immunosuppressive drug treatment.
* Severe kidney failure (estimated glomerular filtration rate < 30 ml/min) or under continuous kidney replacement therapy, hemodialysis, or peritoneal dialysis.
* Immunosuppressed patients (except when the cause is corticosteroid treatment).
* Pregnant or lactating women.
* Patients who plan to become pregnant during the study period or within six months after the end of the study period.
* Participation in another clinical trial with an experimental drug during the last 30 days.
* Pathologies that in medical judgment constitute a contraindication to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change form baseline in Arterial oxygen saturation | up to 25 days
  Pulmonary lesion area will be taken by a chest x-ray or computed axial tomography
Change form baseline in Arterial oxygen saturation | up to 25 days
  Aretrial oxygen saturation will be taken by an oximeter
Days to clinical improvement | up to 25 days
  Number of days of patient discharge

SECONDARY OUTCOMES:
Change Form Baseline in C reactive protein at 25 days | up to 25 days
  Blood samples will be taken on days 1, 3, 7, 15, 20, 25
Change Form Baseline Immune cells: CD3+, CD4+, CD8+, CD16+, CD19+, and CD56+ lymphocytes | up to 25 days
  Blood samples will be taken on days 1, 3, 7, 15, 20, 25
Change Form Baseline in pro-inflammatory cytokines: IL-1β, IL- 2, TNF-α, ITN-γ, IL-4, IL-6, IL-10 | up to 25 days
  Blood samples will be taken on days 1, 3, 7, 15, 20, 25
Change Form Baseline in Immunoglobulins; IgA, IgG, IgM, and IgE. | up to 25 days
  Blood samples will be taken on days 1, 3, 7, 15, 20, 25

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Lic Adolfo Lopez Mateos, Mexico City, Ciudad de Mexico CDMX (Mexico City), Mexico

IPD SHARING:
Plan to Share IPD: No